CLINICAL TRIAL: NCT04157712
Title: A Phase I, Single Centre, Double-Blind, Placebo-Controlled Study of the Safety, Tolerability and Pharmacokinetics in Plasma and Urine of Multiple Ascending Doses of ALZ-801 in Healthy Elderly Subjects
Brief Title: Multiple Ascending Dose Study of ALZ-801
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alzheon Inc. (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ALZ-801-103
Record Dates: First submitted 2019-11-04; First posted 2019-11-08 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — ALZ-801

STUDY DESIGN:
Intervention Model Description: double blind, placebo controlled, matching placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double blind, placebo controlled, matching placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort A Capsule - Fasted (Experimental): ALZ-801 171 mg or matching placebo once daily Day 1, ALZ-801 171 mg or matching placebo twice daily Days 2-7, ALZ-801 256.5 mg or matching placebo once daily Days 8-14
  Interventions: Drug: ALZ-801 or matching placebo
- Cohort B Capsule - Fasted (Experimental): ALZ-801 256.5 mg or matching placebo once daily Day 1, ALZ-801 256.5 or matching placebo mg twice daily Days 2-7, ALZ-801 340 mg or matching placebo once daily Days 8-14
  Interventions: Drug: ALZ-801 or matching placebo
- Cohort C Capsule - Fed (Experimental): ALZ-801 256.5 mg or matching placebo once daily Day 1, ALZ-801 256.5 mg or matching placebo twice daily Days 2-7, ALZ-801 340 mg or matching placebo twice daily Days 8-13, ALZ-801 340 mg or matching placebo once daily Day 14
  Interventions: Drug: ALZ-801 or matching placebo
- Cohort D Tablet - Fed (Experimental): ALZ-801 265 mg or matching placebo once daily Day 1, ALZ-801 265 mg or matching placebo twice daily Days 2-6, ALZ-801 265 mg or matching placebo once daily Day 7
  Interventions: Drug: ALZ-801 or matching placebo

INTERVENTIONS:
Drug: ALZ-801 or matching placebo

SUMMARY:
Phase I, single-center, double-blind, randomized, placebo-controlled, parallel-group study of the safety, tolerability, and pharmacokinetics (PK) in plasma and urine, of multiple ascending doses of ALZ-801 (capsule, Part 1; prototype tablet Part 2) and the primary metabolite in healthy male or female subjects.

DETAILED DESCRIPTION:
The study was conducted in two parts:

Part 1 Primary objective: To evaluate the safety, tolerability, and pharmacokinetics, of multiple doses of ALZ-801 capsule formulation in healthy elderly subjects.

Methodology: Phase I, single center, in-patient and out-patient, double-blind, randomized, placebo-controlled, parallel-group study of the safety, tolerability and pharmacokinetics (PK) in plasma and urine of multiple ascending doses of ALZ-801 in healthy male or female subjects aged 50 to 75 years, inclusive. A total of 36 subjects were enrolled into 3 successive cohorts (A, B, C with 12 subjects per cohort) and randomized in a 3:1 ratio to receive treatment with ALZ-801 capsules (9 subjects) or placebo capsules (3 subjects) for 2 weeks. Progression to the next cohort was permitted after review of safety and available PK data suggested that it was safe to do so. Subjects were confined to the clinical unit for the first day of dosing (Day 1 and for Days 7 through 14). Subjects took investigational drug at home for Days 2 through 6).

Cohorts A was dosed in the fasted state and evaluated 171 mg ALZ-801 or placebo QD for 1 day, followed by 171 mg ALZ-801 or placebo BID for 6 days and 256.5 mg or placebo QD for 7 days.

Cohort B was dosed in the fasted state and evaluated 256.5 mg ALZ-801 or placebo QD for 1 day, followed by 256.5 mg ALZ-801 or placebo BID for 6 days and 340 mg or placebo QD for 7 days.

Cohort C was dosed in the fed state and evaluated 256.5 mg ALZ-801 or placebo QD for 1 day, followed by 256.5 mg ALZ-801 or placebo BID for 6 days, then 340 mg or placebo BID for 6 days and 340 mg or placebo QD for 1 day.

Part 2 Primary objective: To evaluate the safety, tolerability, and pharmacokinetics, of multiple doses of prototype ALZ-801 tablet formulation in healthy elderly subjects.

Methodology: Phase I, single center, in-patient and out-patient, double-blind, randomized, placebo-controlled, parallel-group study of the safety, tolerability and pharmacokinetics (PK) in plasma and urine of multiple ascending doses of ALZ-801 in healthy male or female subjects aged 60 to 75 years, inclusive. A total of 12 subjects were enrolled into one cohort (D) and randomized in a 3:1 ratio to receive treatment with ALZ-801 tablets (9 subjects) or placebo capsules (3 subjects) for 1 week.

Cohort D was dosed in the fed state and evaluated 265 mg ALZ-801 or placebo QD for 1 day, followed by 265 mg ALZ-801 prototype tablet or placebo BID for 5 days, 265 mg or placebo QD for 1 day.

For all subjects in the study blood and urine samples for the determination of concentrations of ALZ-801, and its metabolites, were collected for up to 24 h after the first dose of medication on Day1; and for up to 48 hours after the last dose of medication on Day 7 (Cohort D) or Day 14 (Cohorts A, B and C). All subjects had blood samples and safety assessment at 72 and 96 hours after the final dose of medication. All subjects returned for a post treatment follow-up 7-10 days after the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males, and females
* Age: 50-75 years, Part 1; 60-75 years Part 2
* Females must be of non-childbearing potential
* Body Mass Index 18-35 kg/m squared;
* Vital signs normal for age: BP 90-160/40-90 mmHg; HR 50 to 90 bpm)
* No clinically significant electrocardiogram readings

Exclusion Criteria:

* Body weight < 50 kg
* History of any drug or alcohol abuse in the past 2 years
* Subjects known to have a creatinine clearance of <60 mL/min
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
* History of clinically significant cardiovascular, pulmonary, chronic respiratory, renal, hepatic, GI, immunologic, endocrine, neurologic, psychiatric or thromboembolic disease
* History of metabolic disturbances;

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-09-26 (Actual); Primary Completion 2016-07-04 (Actual); Study Completion 2016-07-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Duration of dosing: 14 days for Part 1; 7 days for Part 2
  Incidence and nature of adverse events (AEs) and serious adverse events (SAEs). Assessments reported as AEs or SAEs include physical examination, clinical laboratory tests, and 12-lead electrocardiogram (ECG) findings
Cmax for ALZ-801 and tramiprosate | Days 1, 7 and 14
  Maximum concentration after dosing [Cmax] measured as ng/ml
Tmax for ALZ-801 and tramiprosate | Days 1, 7 and 14
  Time to reach Cmax [Tmax] measured in hours (h) after dosing
AUC for ALZ-801 and tramiprosate | Days 1, 7 and 14
  AUC from time zero to time t (AUCt)
t1/2 for ALZ-801 and tramiprosate | Days 1, 7, 14
  Elimination half-life (t1/2) measured in hours after dosing
Renal clearance of ALZ-801 and tramiprosate | Days 1, 7 and 14
  Clearance (CLr) measured in mL/min

CONTACTS AND LOCATIONS:
Overall Officials: Pui Leung, MD, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hey JA, Yu JY, Versavel M, Abushakra S, Kocis P, Power A, Kaplan PL, Amedio J, Tolar M. Clinical Pharmacokinetics and Safety of ALZ-801, a Novel Prodrug of Tramiprosate in Development for the Treatment of Alzheimer's Disease. Clin Pharmacokinet. 2018 Mar;57(3):315-333. doi: 10.1007/s40262-017-0608-3. PMID 29063518